CLINICAL TRIAL: NCT04274075
Title: A Phase 1, Open-Label, Single-Dose, Randomized, Three-Period Crossover Study to Evaluate the Relative Bioavailability and Food Effect of GDC-9545 in Healthy Female Subjects of Non-Childbearing Potential
Brief Title: Evaluation of the Relative Bioavailability and Food Effect of GDC-9545 in Healthy Females of Non-Childbearing Potential
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GP42006
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — giredestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- GDC-9545 Treatment Sequence A, B, and C (Experimental): Participants randomized to this arm will receive one dose of GDC-9545 at the start of each of three periods according to the treatment sequence A, B, and C (refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
  Interventions: Drug: GDC-9545 Tablet, Fasted: Treatment A; Drug: GDC-9545 Capsule, Fasted: Treatment B; Drug: GDC-9545 Capsule, Fed: Treatment C
- GDC-9545 Treatment Sequence B, C, and A (Experimental): Participants randomized to this arm will receive one dose of GDC-9545 at the start of each of three periods according to the treatment sequence B, C, and A (refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
  Interventions: Drug: GDC-9545 Tablet, Fasted: Treatment A; Drug: GDC-9545 Capsule, Fasted: Treatment B; Drug: GDC-9545 Capsule, Fed: Treatment C
- GDC-9545 Treatment Sequence C, A, and B (Experimental): Participants randomized to this arm will receive one dose of GDC-9545 at the start of each of three periods according to the treatment sequence C, A, and B (refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
  Interventions: Drug: GDC-9545 Tablet, Fasted: Treatment A; Drug: GDC-9545 Capsule, Fasted: Treatment B; Drug: GDC-9545 Capsule, Fed: Treatment C
- GDC-9545 Treatment Sequence A, C, and B (Experimental): Participants randomized to this arm will receive one dose of GDC-9545 at the start of each of three periods according to the treatment sequence A, C, and B (refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
  Interventions: Drug: GDC-9545 Tablet, Fasted: Treatment A; Drug: GDC-9545 Capsule, Fasted: Treatment B; Drug: GDC-9545 Capsule, Fed: Treatment C
- GDC-9545 Treatment Sequence B, A, and C (Experimental): Participants randomized to this arm will receive one dose of GDC-9545 at the start of each of three periods according to the treatment sequence B, A, and C (refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
  Interventions: Drug: GDC-9545 Tablet, Fasted: Treatment A; Drug: GDC-9545 Capsule, Fasted: Treatment B; Drug: GDC-9545 Capsule, Fed: Treatment C
- GDC-9545 Treatment Sequence C, B, and A (Experimental): Participants randomized to this arm will receive one dose of GDC-9545 at the start of each of three periods according to the treatment sequence C, B, and A (refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
  Interventions: Drug: GDC-9545 Tablet, Fasted: Treatment A; Drug: GDC-9545 Capsule, Fasted: Treatment B; Drug: GDC-9545 Capsule, Fed: Treatment C

INTERVENTIONS:
Drug: GDC-9545 Tablet, Fasted: Treatment A — One dose of the GDC-9545 Phase 1 reference tablet formulation (three 10-mg tablets) administered orally with approximately 240 mL room temperature water after at least an 8-hour fast.
  Other Names: Giredestrant; RO7197597; RG6171
Drug: GDC-9545 Capsule, Fasted: Treatment B — One dose of the GDC-9545 Phase 3 capsule formulation (one 30-mg capsule) administered orally with approximately 240 mL room temperature water after at least an 8-hour fast.
  Other Names: Giredestrant; RO7197597; RG6171
Drug: GDC-9545 Capsule, Fed: Treatment C — One dose of the GDC-9545 Phase 3 capsule formulation (one 30-mg capsule) administered orally with approximately 240 mL room temperature water within 30 minutes of eating a high-fat meal.
  Other Names: Giredestrant; RO7197597; RG6171

SUMMARY:
This study will be an open-label, randomized, three-period, six-sequence crossover study of GDC-9545 administered to healthy females of non-childbearing potential to determine the relative bioavailability of the Phase 3 capsule formulation to the Phase 1 tablet formulation in the fasted state and the effect of food on the Phase 3 capsule formulation.

ELIGIBILITY:
Inclusion Criteria:

* Females of non-childbearing potential including non-pregnant, non-lactating, and either postmenopausal or surgically sterile for at least 90 days prior to screening, as defined in the protocol
* Body mass index (BMI) from 18.5 to 30.0 kilograms per square metre of body surface area (kg/m^2) at screening
* In good health, determined by no clinically significant findings from medical history, 12-lead ECG, or vital signs
* Clinical laboratory evaluations within the reference range for the test laboratory, unless deemed not clinically significant by the investigator
* Negative test for selected drugs of abuse at Screening (does not include alcohol) and at Check-in (Day -1) for Period 1 (does include alcohol)
* Negative hepatitis panel (hepatitis B surface antigen and hepatitis C virus antibody) and negative human immunodeficiency virus (HIV) antibody screens
* Subject must receive an explanation of the mandatory Research Biosample Repository (RBR) component of the study and be able to comprehend and willing to sign an Informed Consent Form (ICF)

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal (GI), neurological, or psychiatric disorder (as determined by the investigator)
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator
* History of allergy to GDC-9545 or any of its excipients
* History of stomach or intestinal surgery (including cholecystectomy) or resection that would potentially alter absorption and/or excretion of orally administered drugs (except that appendectomy and hernia repair will be allowed)
* History or presence of an abnormal ECG that, in the investigator's opinion, is clinically significant including complete left bundle branch block; right bundle branch block; first-, second-, or third-degree heart block; sick sinus syndrome; or evidence of prior myocardial infarction
* Having a QTc interval greater than (>)470 milliseconds (msec), PR interval >210 msec, or QRS complex >120 msec
* Confirmed (e.g., 2 consecutive measurements) baseline heart rate ≤50 beats per minute (bpm) prior to enrollment
* History of alcoholism or drug addiction within 1 year prior to Check-in (Day -1) of Period 1
* The use of tobacco- or nicotine-containing products within 6 months prior to Check-in (Day -1) of Period 1
* History of active or latent tuberculosis (TB), regardless of treatment history
* History of previous use of tamoxifen, aromatase inhibitors, or any other endocrine agent for the treatment of breast cancer
* The use of hormone replacement therapy or selective ER modulators (SERMs; e.g., raloxifene) within 1 year prior to Check-in (Day -1) of Period 1
* The use of oral antibiotics within 4 weeks or intravenous antibiotics within 8 weeks prior to Check-in (Day -1) of Period 1
* The use or intent to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to Check-in (Day -1) of Period 1
* The participation in any other investigational study drug trial in which receipt of an investigational study drug occurred within 5 half-lives or 30 days, whichever is longer, prior to Check-in (Day -1) of Period 1
* The use of drugs of abuse (including opioids) within 4 weeks of Screening
* The use of any prescription medications/products within 14 days prior to Check-in (Day -1) of Period 1, unless deemed acceptable by the investigator
* The use of any over-the-counter, non-prescription preparations (including vitamins; minerals; and phytotherapeutic-, herbal-, and plant-derived preparations) within 7 days prior to Check-in (Day -1) of Period 1, unless deemed acceptable by the investigator
* The use of poppy seed-containing foods or beverages within 7 days prior to Check-in (Day -1) of Period 1, unless deemed acceptable by the investigator
* The use of alcohol- or caffeine-containing foods or beverages within 72 hours prior to Check-in (Day -1) of Period 1, unless deemed acceptable by the investigator
* Not refraining from strenuous exercise from 7 days prior to Check-in (Day -1) of Period 1
* The need to follow a special diet and unable to consume the high-fat meal
* Poor peripheral venous access
* History of malignancy, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, or Stage I uterine cancer (must be cancer-free for at least 5 years)
* Donation of blood from 90 days prior to Screening through Follow-up, inclusive, or of plasma from 2 weeks prior to Screening
* Receipt of blood products within 2 months prior to Check-in (Day -1) of Period 1
* Any acute or chronic condition that, in the opinion of the investigator, would limit the subject's ability to complete and/or participate in this clinical study
* In the opinion of the investigator or Sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-04-16 (Actual); Study Completion 2020-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Covance Research Unit - Daytona, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/).
  For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

RESULTS

PARTICIPANT FLOW:
Groups:
- GDC-9545 Treatment Sequence A, B, and C: Participants randomized to this arm received one dose of GDC-9545 at the start (Day 1) of each of three treatment periods according to the treatment cross-over sequence A, B, and C (please refer to the intervention descriptions). The washout period between doses was a minimum of 10 days.
- GDC-9545 Treatment Sequence B, C, and A: Participants randomized to this arm received one dose of GDC-9545 at the start (Day 1) of each of three treatment periods according to the treatment cross-over sequence B, C, and A (please refer to the intervention descriptions). The washout period between doses was a minimum of 10 days.
- GDC-9545 Treatment Sequence C, A, and B: Participants randomized to this arm received one dose of GDC-9545 at the start (Day 1) of each of three treatment periods according to the treatment cross-over sequence C, A, and B (please refer to the intervention descriptions). The washout period between doses was a minimum of 10 days.
- GDC-9545 Treatment Sequence A, C, and B: Participants randomized to this arm received one dose of GDC-9545 at the start (Day 1) of each of three treatment periods according to the treatment cross-over sequence A, C, and B (please refer to the intervention descriptions). The washout period between doses was a minimum of 10 days.
- GDC-9545 Treatment Sequence B, A, and C: Participants randomized to this arm received one dose of GDC-9545 at the start (Day 1) of each of three treatment periods according to the treatment cross-over sequence B, A, and C (please refer to the intervention descriptions). The washout period between doses was a minimum of 10 days.
- GDC-9545 Treatment Sequence C, B, and A: Participants randomized to this arm received one dose of GDC-9545 at the start (Day 1) of each of three treatment periods according to the treatment cross-over sequence C, B, and A (please refer to the intervention descriptions). The washout period between doses will be a minimum of 10 days.
Period: Overall Study
Arm/Group | GDC-9545 Treatment Sequence A, B, and C | GDC-9545 Treatment Sequence B, C, and A | GDC-9545 Treatment Sequence C, A, and B | GDC-9545 Treatment Sequence A, C, and B | GDC-9545 Treatment Sequence B, A, and C | GDC-9545 Treatment Sequence C, B, and A
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed Treatment Period 1 (9 Days) | 3 | 3 | 3 | 3 | 3 | 3
Completed Treatment Period 2 (9 Days) | 3 | 3 | 3 | 3 | 3 | 3
Completed Treatment Period 3 (9 Days) | 3 | 3 | 3 | 3 | 3 | 3
Completed Follow-up Visit (The follow-up visit took place 12 to 14 days after the last dose of study drug.) | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GDC-9545 Treatment Sequence A, B, and C | GDC-9545 Treatment Sequence B, C, and A | GDC-9545 Treatment Sequence C, A, and B | GDC-9545 Treatment Sequence A, C, and B | GDC-9545 Treatment Sequence B, A, and C | GDC-9545 Treatment Sequence C, B, and A | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.0 (4.4) | 55.0 (5.2) | 48.3 (8.1) | 54.0 (9.5) | 56.3 (5.9) | 53.7 (4.9) | 53.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 3 | 3 | 18
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 1 | 2 | 3 | 11
  Not Hispanic or Latino | 1 | 2 | 1 | 2 | 1 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 3 | 3 | 3 | 3 | 18

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of GDC-9545
Description: The pharmacokinetics (PK) parameters were determined where possible from the plasma concentrations of GDC-9545 using non-compartmental methods performed using Phoenix WinNonlin. The PK parameters Cmax, AUC0-t, and AUC0-∞ for GDC-9545 were analyzed to evaluate the relative bioavailability of GDC-9545 as a Phase 3 capsule formulation compared to a Phase 1 tablet formulation under fasted conditions (Treatment B vs. Treatment A) and to assess the food effect on GDC-9545 PK for a Phase 3 capsule formulation (Treatment C vs. Treatment B). The mixed-effect analysis of variance model for three-period crossover design was used for formulation comparison and fasted state and fed state comparison of capsule. The model included sequence, formulation, and period as fixed effects and a random effect for subject within sequence. An unstructured covariance structure was to be used; however, if it failed to converge, an alternative covariance structure may have been applied.
Time Frame: Pre-dose (0 hour) and post-dose at 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, and 12 hours on Day 1 and post-dose once a day on Days 2 to 8 of Periods 1-3 (up to 27 days)
Population: Pharmacokinetics (PK) Population: all participants who received at least one dose of study drug and had at least one evaluable postdose PK sample, with participants grouped according to the treatment received.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Groups:
- GDC-9545 Tablet, Fasted: Treatment A: This analysis population consisted of all participants who were enrolled in the study, regardless of the treatment sequence arm to which they were randomized, and received one dose of GDC-9545 Treatment A. Treatment A consisted of one dose of the GDC-9545 Phase 1 reference tablet formulation (three 10-mg tablets) administered orally with approximately 240 mL room temperature water after at least an 8-hour fast.
- GDC-9545 Capsule, Fasted: Treatment B: This analysis population consisted of all participants who were enrolled in the study, regardless of the treatment sequence arm to which they were randomized, and received one dose of GDC-9545 Treatment B. Treatment B consisted of one dose of the GDC-9545 Phase 3 capsule formulation (one 30-mg capsule) administered orally with approximately 240 mL room temperature water after at least an 8-hour fast.
- GDC-9545 Capsule, Fed: Treatment C: This analysis population consisted of all participants who were enrolled in the study, regardless of the treatment sequence arm to which they were randomized, and received one dose of GDC-9545 Treatment C. Treatment C consisted of one dose of the GDC-9545 Phase 3 capsule formulation (one 30-mg capsule) administered orally with approximately 240 mL room temperature water within 30 minutes of eating a high-fat meal.
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
nanograms per millilitre (ng/mL) | 126 (29.6) | 129 (27.7) | 102 (27.3)
Statistical Analysis 1: Comparison: GDC-9545 Tablet, Fasted: Treatment A vs GDC-9545 Capsule, Fasted: Treatment B; The sample size chosen for this study was based upon precedent set by other PK studies of similar nature and was not based on power calculations; Test type: Other; Geometric Mean Ratio = 1.03, 90% CI 2-sided [0.945 to 1.12] — The geometric mean ratio was calculated as Treatment B versus Treatment A
Statistical Analysis 2: Comparison: GDC-9545 Capsule, Fasted: Treatment B vs GDC-9545 Capsule, Fed: Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean Ratio = 0.790, 90% CI 2-sided [0.726 to 0.859] — The geometric mean ratio was calculated as Treatment C versus Treatment B

2. Primary Outcome: Time to Maximum Observed Plasma Concentration (Tmax) of GDC-9545
Description: The pharmacokinetics (PK) parameters were determined where possible from the plasma concentrations of GDC-9545 using non-compartmental methods performed using Phoenix WinNonlin. The parameter tmax was analyzed nonparametrically using the Wilcoxon signed-rank test. The median difference between the test and reference investigational products (GDC-9545 Phase 3 capsule formulation compared to a Phase 1 tablet formulation under fasted conditions [Treatment B vs. Treatment A] and the food effect on GDC-9545 PK for a Phase 3 capsule formulation [Treatment C vs. Treatment B]) and the corresponding 90% confidence interval were calculated.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Hours | 2.25 [1.00 to 5.00] | 2.28 [1.50 to 5.00] | 5.00 [3.00 to 6.00]
Statistical Analysis 1: Comparison: GDC-9545 Tablet, Fasted: Treatment A vs GDC-9545 Capsule, Fasted: Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other; Median Difference (Net) = 0.525, 90% CI 2-sided [-0.225 to 1.50] — The Hodges-Lehmann estimate of median difference was calculated as Treatment B versus Treatment A
Statistical Analysis 2: Comparison: GDC-9545 Capsule, Fasted: Treatment B vs GDC-9545 Capsule, Fed: Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Median Difference (Net) = 1.98, 90% CI 2-sided [1.26 to 2.45] — The Hodges-Lehmann estimate of median difference was calculated as Treatment C versus Treatment B

3. Primary Outcome: Time of Last Quantifiable Plasma Concentration (Tlast) of GDC-9545
Description: The pharmacokinetics parameters were determined where possible from the plasma concentrations of GDC-9545 using non-compartmental methods performed using Phoenix WinNonlin.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Hours | 168 [168 to 168] | 168 [168 to 168] | 168 [168 to 168]

4. Primary Outcome: Time to First Quantifiable Plasma Concentration (Tlag) of GDC-9545
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: Hours
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Hours | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 1.00]

5. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Hour 0 to the Last Measurable Concentration (AUC0-t) of GDC-9545
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*ng/mL
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Hours*ng/mL | 3710 (31.8) | 3600 (29.8) | 3310 (27.6)
Statistical Analysis 1: Comparison: GDC-9545 Tablet, Fasted: Treatment A vs GDC-9545 Capsule, Fasted: Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean Ratio = 0.971, 90% CI 2-sided [0.903 to 1.04] — The geometric mean ratio was calculated as Treatment B versus Treatment A
Statistical Analysis 2: Comparison: GDC-9545 Capsule, Fasted: Treatment B vs GDC-9545 Capsule, Fed: Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean Ratio = 0.919, 90% CI 2-sided [0.855 to 0.988] — The geometric mean ratio was calculated as Treatment C versus Treatment B

6. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Hour 0 Extrapolated to Infinity (AUC0-∞) of GDC-9545
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours*ng/mL
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Hours*ng/mL | 3860 (32.6) | 3770 (30.8) | 3460 (28.1)
Statistical Analysis 1: Comparison: GDC-9545 Tablet, Fasted: Treatment A vs GDC-9545 Capsule, Fasted: Treatment B; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean Ratio = 0.975, 90% CI 2-sided [0.908 to 1.05] — The geometric mean ratio was calculated as Treatment B versus Treatment A
Statistical Analysis 2: Comparison: GDC-9545 Capsule, Fasted: Treatment B vs GDC-9545 Capsule, Fed: Treatment C; [analysis description as in outcome 1, analysis 1]; Test type: Other; Geometric Mean Ratio = 0.918, 90% CI 2-sided [0.856 to 0.985] — The geometric mean ratio was calculated as Treatment C versus Treatment B

7. Primary Outcome: Percentage of Area Under the Plasma Concentration-Time Curve (AUC) That is Due to Extrapolation From Last Measurable Concentration to Infinity (%AUCextrap) of GDC-9545
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of AUC
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Percentage of AUC | 3.40 (58.5) | 3.87 (49.8) | 3.78 (48.9)

8. Primary Outcome: Apparent Terminal Elimination Rate Constant (λz) of GDC-9545
Description: The pharmacokinetics parameters were determined where possible from the plasma concentrations of GDC-9545 using non-compartmental methods performed using Phoenix WinNonlin. The apparent terminal elimination rate constant (λz) is the magnitude of the slope of the linear regression of the log concentration versus time profile during the terminal phase.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Elimination rate per hour (/h)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Elimination rate per hour (/h) | 0.0196 (15.7) | 0.0185 (15.5) | 0.0188 (14.4)

9. Primary Outcome: Apparent Terminal Elimination Half-Life (t1/2) of GDC-9545
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Hours | 35.4 (15.7) | 37.4 (15.5) | 36.9 (14.4)

10. Primary Outcome: Apparent Total Clearance (CL/F) of GDC-9545
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour (L/h)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Litres per hour (L/h) | 7.76 (32.6) | 7.97 (30.8) | 8.68 (28.1)

11. Primary Outcome: Apparent Volume of Distribution During the Terminal Elimination Phase (Vz/F) of GDC-9545
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres (L)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Litres (L) | 397 (29.8) | 430 (26.5) | 462 (29.8)

12. Secondary Outcome: Number of Participants Who Experienced at Least One Adverse Event by Severity, According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI-CTCAE v5.0)
Description: The investigator sought information on adverse events (AEs) at each contact with a participant. All AEs, whether reported by the participant or noted by study personnel, were recorded. All AEs were assigned a severity grade (from 1 to 5) using the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0). Severity refers to the intensity of an AE. The following is the severity grading scale used for AEs that are not specifically listed in the NCI-CTCAE: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening; and Grade 5 is death related to an AE.
Time Frame: From first dose of study drug until 14 days after the last dose of study drug (up to 41 days)
Population: Safety Population: all participants who received at least one dose of study drug, with participants grouped according to the treatment received.
Measure: Count of Participants; unit: Participants
Groups:
- Overall: Any GDC-9545 Treatment (A, B, or C): This analysis population consisted of all participants who were enrolled in the study, regardless of the treatment sequence arm to which they were randomized, and received at least one dose of any study drug (GDC-9545 Treatments A, B, or C).
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C | Overall: Any GDC-9545 Treatment (A, B, or C)
Number analyzed (Participants) | 18 | 18 | 18 | 18
Participants
  Any Adverse Event (AE), Any Grade | 2 | 2 | 3 | 5
  AE by Initial Severity, Grade 1 | 2 | 2 | 2 | 4
  AE by Initial Severity, Grade 2 | 0 | 0 | 1 | 1
  AE by Initial Severity, Grade 3 | 0 | 0 | 0 | 0
  AE by Initial Severity, Grade 4 | 0 | 0 | 0 | 0
  AE by Initial Severity, Grade 5 | 0 | 0 | 0 | 0
  AE by Most Extreme Severity, Grade 1 | 2 | 2 | 2 | 4
  AE by Most Extreme Severity, Grade 2 | 0 | 0 | 1 | 1
  AE by Most Extreme Severity, Grade 3 | 0 | 0 | 0 | 0
  AE by Most Extreme Severity, Grade 4 | 0 | 0 | 0 | 0
  AE by Most Extreme Severity, Grade 5 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Chemistry, Hematology, and Urinalysis Laboratory Tests
Description: Participants provided blood and urine samples at the specified timepoints for laboratory analysis of clinical chemistry, hematology, and urinalysis parameters (please refer to Appendix A of the protocol for a complete list of parameters). Any of the laboratory test results that were outside of the reference range were considered abnormalities. Not every laboratory abnormality qualified as an adverse event (AE). A laboratory test result was reported as an AE if it met any of the following criteria: was accompanied by clinical symptoms; resulted in a change in study treatment; resulted in a medical intervention or a change in concomitant therapy; or was clinically significant in the investigator's judgment. All AEs were assigned a severity grade (from 1 to 5) using the NCI-CTCAE v5.0; for AEs not specifically listed in the NCI-CTCAE: Grade 1 is mild; Grade 2 is moderate; Grade 3 is severe or medically significant; Grade 4 is life-threatening; and Grade 5 is death related to an AE.
Time Frame: Baseline, Days 2 and 8 of Period 1-3, and 12-14 days after last dose (up to 34 days)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Participants | 0 | 0 | 1

14. Secondary Outcome: Change From Baseline in Systolic Blood Pressure Over Time
Description: Vital signs (including oral temperature, respiratory rate, and supine blood pressure and pulse rate) were obtained at the specified timepoints. Supine blood pressure was obtained after the participant had been supine for at least 5 minutes. When vital signs were scheduled at the same time as blood draws, the blood draws were obtained at the scheduled timepoint, and the vital signs were obtained as close to the scheduled blood draw as possible, but prior to the blood draw. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The normal reference range for supine systolic blood pressure was 90-140 millimetres of mercury (mmHg).
Time Frame: Baseline and post-dose on Days 1 to 8 of Periods 1-3 (up to 27 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
millimetres of mercury (mmHg)
  Baseline (BL) - Value at Visit | 104.5 (12.03) | 103.1 (8.73) | 102.6 (9.28)
  Change from BL at Day 1 | -1.7 (7.17) | 0.7 (10.50) | -3.8 (7.33)
  Change from BL at Day 2 | -5.9 (6.93) | -4.0 (9.39) | -1.2 (7.77)
  Change from BL at Day 3 | -3.7 (7.46) | -1.8 (8.71) | -1.1 (8.39)
  Change from BL at Day 4 | -2.8 (7.56) | -3.2 (7.61) | -2.6 (9.65)
  Change from BL at Day 5 | -4.9 (7.03) | -2.6 (6.46) | -3.8 (6.71)
  Change from BL at Day 6 | -5.3 (8.94) | -1.8 (6.39) | -0.6 (8.95)
  Change from BL at Day 7 | -5.2 (8.19) | -3.3 (7.31) | -2.9 (8.12)
  Change from BL at Day 8 | -3.4 (9.23) | -0.4 (6.68) | -2.3 (6.28)

15. Secondary Outcome: Change From Baseline in Diastolic Blood Pressure Over Time
Description: Vital signs (including oral temperature, respiratory rate, and supine blood pressure and pulse rate) were obtained at the specified timepoints. Supine blood pressure was obtained after the participant had been supine for at least 5 minutes. When vital signs were scheduled at the same time as blood draws, the blood draws were obtained at the scheduled timepoint, and the vital signs were obtained as close to the scheduled blood draw as possible, but prior to the blood draw. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The normal reference range for supine diastolic blood pressure was 50-90 mmHg.
Time Frame: Baseline and Days 1 to 8 of Periods 1-3 (up to 27 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: millimetres of mercury (mmHg)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
millimetres of mercury (mmHg)
  Baseline (BL) - Value at Visit | 64.2 (7.86) | 62.5 (8.40) | 62.8 (7.67)
  Change from BL at Day 1 | -2.8 (5.31) | -3.1 (6.73) | -3.3 (6.23)
  Change from BL at Day 2 | -3.2 (6.13) | -2.7 (8.73) | -1.6 (6.64)
  Change from BL at Day 3 | -4.2 (6.96) | 0.2 (7.52) | -1.0 (6.87)
  Change from BL at Day 4 | -2.3 (4.67) | -2.3 (7.50) | -2.3 (6.44)
  Change from BL at Day 5 | -2.8 (7.36) | -0.9 (5.31) | -2.3 (6.82)
  Change from BL at Day 6 | -4.3 (6.13) | -1.8 (6.37) | -0.4 (7.22)
  Change from BL at Day 7 | -3.1 (7.07) | -0.9 (6.10) | -1.8 (6.83)
  Change from BL at Day 8 | -3.1 (6.66) | 0.1 (7.45) | -3.3 (7.39)

16. Secondary Outcome: Change From Baseline in Pulse Rate Over Time
Description: Vital signs (including oral temperature, respiratory rate, and supine blood pressure and pulse rate) were obtained at the specified timepoints. Supine pulse rate was obtained after the participant had been supine for at least 5 minutes. When vital signs were scheduled at the same time as blood draws, the blood draws were obtained at the scheduled timepoint, and the vital signs were obtained as close to the scheduled blood draw as possible, but prior to the blood draw. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The normal reference range for supine pulse rate was 40-100 beats per minute.
Time Frame: Baseline and Days 1 to 8 of Periods 1-3 (up to 27 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Beats per minute
  Baseline (BL) - Value at Visit | 62.2 (7.61) | 62.4 (8.88) | 65.3 (11.00)
  Change from BL at Day 1 | -2.1 (6.27) | -4.1 (7.62) | -1.3 (9.39)
  Change from BL at Day 2 | 1.4 (10.34) | -3.2 (7.65) | -5.4 (7.01)
  Change from BL at Day 3 | -0.6 (5.61) | -4.1 (6.29) | -4.8 (7.73)
  Change from BL at Day 4 | -1.1 (8.08) | -2.2 (9.52) | -5.6 (7.85)
  Change from BL at Day 5 | -1.1 (6.76) | -2.8 (6.67) | -4.7 (9.33)
  Change from BL at Day 6 | -0.2 (7.58) | -0.4 (8.60) | -4.4 (8.56)
  Change from BL at Day 7 | -0.7 (7.10) | -1.4 (5.99) | -5.4 (8.20)
  Change from BL at Day 8 | 1.1 (9.00) | -0.1 (7.19) | -2.6 (6.30)

17. Secondary Outcome: Change From Baseline in Respiratory Rate Over Time
Description: Vital signs (including oral temperature, respiratory rate, and supine blood pressure and pulse rate) were obtained at the specified timepoints. When vital signs were scheduled at the same time as blood draws, the blood draws were obtained at the scheduled timepoint, and the vital signs were obtained as close to the scheduled blood draw as possible, but prior to the blood draw. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The normal reference range for respiratory rate was 10-24 breaths per minute.
Time Frame: Baseline and Days 1 to 8 of Periods 1-3 (up to 27 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Breaths per minute
  Baseline (BL) - Value at Visit | 15.6 (1.76) | 15.6 (1.89) | 15.6 (2.01)
  Change from BL at Day 1 | 1.6 (2.53) | 1.2 (1.96) | 2.0 (3.14)
  Change from BL at Day 2 | -0.6 (2.90) | -0.7 (3.07) | -0.8 (2.29)
  Change from BL at Day 3 | -0.4 (2.71) | -0.6 (3.55) | -0.6 (3.35)
  Change from BL at Day 4: number analyzed (Participants) | 18 | 17 | 18
  Change from BL at Day 4 | 0.1 (2.00) | 0.2 (2.54) | -0.3 (2.68)
  Change from BL at Day 5 | 0.8 (3.60) | 0.1 (2.70) | 1.0 (2.93)
  Change from BL at Day 6 | 0.0 (2.74) | 0.2 (2.37) | -0.6 (3.20)
  Change from BL at Day 7 | -0.4 (3.26) | -1.0 (3.31) | -0.8 (3.15)
  Change from BL at Day 8 | -0.9 (1.97) | -1.1 (2.30) | -1.0 (2.40)

18. Secondary Outcome: Change From Baseline in Oral Body Temperature Over Time
Description: Vital signs (including oral temperature, respiratory rate, and supine blood pressure and pulse rate) were obtained at the specified timepoints. When vital signs were scheduled at the same time as blood draws, the blood draws were obtained at the scheduled timepoint, and the vital signs were obtained as close to the scheduled blood draw as possible, but prior to the blood draw. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The normal reference range for oral body temperature was 35.5-37.8 degrees Celsius (C).
Time Frame: Baseline and Days 1 to 8 of Periods 1-3 (up to 27 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: degrees Celsius (C)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
degrees Celsius (C)
  Baseline (BL) - Value at Visit | 36.65 (0.142) | 36.64 (0.115) | 36.72 (0.129)
  Change from BL at Day 1 | 0.06 (0.129) | 0.00 (0.124) | 0.04 (0.195)
  Change from BL at Day 2 | 0.12 (0.183) | 0.07 (0.149) | 0.00 (0.150)
  Change from BL at Day 3 | 0.12 (0.140) | 0.11 (0.229) | 0.03 (0.119)
  Change from BL at Day 4 | 0.08 (0.182) | 0.09 (0.189) | 0.03 (0.146)
  Change from BL at Day 5 | 0.12 (0.163) | 0.11 (0.184) | 0.03 (0.161)
  Change from BL at Day 6 | 0.08 (0.150) | 0.11 (0.195) | 0.03 (0.137)
  Change from BL at Day 7 | 0.08 (0.158) | 0.10 (0.128) | 0.06 (0.138)
  Change from BL at Day 8 | 0.12 (0.202) | 0.13 (0.124) | 0.01 (0.135)

19. Secondary Outcome: Change From Baseline in Duration of PR, RR, QRS, QT, QTcB, and QTcF Intervals Over Time, as Measured by Electrocardiogram
Description: A single 12-lead electrocardiogram (ECG) was obtained at the specified timepoints. To minimize variability in autonomic tone and heart rate, participants rested quietly and in a supine position for at least 5 minutes prior to recording the ECG. Blood draws, other procedures, activity, and environmental distractions (e.g., television, radio, conversation) were to be avoided during the pre-ECG resting period and between ECG recordings to minimize variability due to the effects of activity and stress on cardiac electrophysiology. Whenever possible, ECG tracings for each participant were to be obtained from the same type of machine throughout the study. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The following are the normal reference ranges for ECG interval durations in milliseconds (msec): PR [120-210 msec]; QRS [upper limit: <120 msec]; QT, QTcB, and QTcF [upper limit: <470 msec].
Time Frame: Baseline, and pre-dose and 4 hours post-dose on Day 1, and post-dose on Days 2, and 8 of Periods 1-3 (up to 27 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
milliseconds (msec)
  PR: Baseline (BL) - Value at Visit | 170.2 (15.38) | 171.5 (13.87) | 165.8 (17.39)
  PR: Change from BL at Day 1 | -3.6 (5.80) | -6.1 (7.37) | -2.7 (13.46)
  PR: Change from BL at Day 2 | -3.9 (10.65) | -4.8 (11.93) | 4.4 (8.32)
  PR: Change from BL at Day 8 | -2.1 (9.32) | -4.4 (9.43) | -1.0 (10.58)
  RR: Baseline (BL) - Value at Visit | 966.7 (115.12) | 986.8 (106.40) | 971.6 (131.35)
  RR: Change from BL at Day 1 | 43.9 (64.10) | 64.6 (113.36) | -6.0 (134.23)
  RR: Change from BL at Day 2 | 19.6 (88.42) | 55.0 (97.58) | 66.7 (89.61)
  RR: Change from BL at Day 8 | -1.3 (74.84) | -12.6 (71.04) | 9.9 (89.01)
  QRS: Baseline (BL) - Value at Visit | 87.4 (8.79) | 88.9 (7.59) | 89.4 (8.93)
  QRS: Change from BL at Day 1 | -0.1 (5.01) | 0.6 (3.66) | -4.4 (8.65)
  QRS: Change from BL at Day 2 | 0.7 (5.01) | -0.7 (5.28) | -2.1 (5.78)
  QRS: Change from BL at Day 8 | -0.6 (5.18) | -1.5 (4.93) | -1.7 (4.36)
  QT: Baseline (BL) - Value at Visit | 414.7 (21.01) | 416.5 (18.51) | 411.9 (25.22)
  QT: Change from BL at Day 1 | 5.9 (11.93) | 11.4 (15.44) | -9.7 (18.23)
  QT: Change from BL at Day 2 | 0.5 (16.45) | 5.7 (16.12) | 11.9 (13.27)
  QT: Change from BL at Day 8 | -2.6 (11.78) | -2.8 (10.71) | 1.6 (15.15)
  QTcB: Baseline (BL) - Value at Visit | 422.3 (12.45) | 419.9 (15.40) | 418.7 (12.68)
  QTcB: Change from BL at Day 1 | -3.3 (12.28) | -1.7 (12.72) | -7.9 (17.39)
  QTcB: Change from BL at Day 2 | -3.4 (11.72) | -5.4 (10.99) | -2.1 (12.89)
  QTcB: Change from BL at Day 8 | -2.4 (12.46) | -0.2 (11.90) | -0.6 (10.54)
  QTcF: Baseline (BL) - Value at Visit | 419.5 (11.10) | 418.3 (12.85) | 415.9 (11.91)
  QTcF: Change from BL at Day 1 | -0.2 (10.38) | 2.8 (8.50) | -8.5 (12.22)
  QTcF: Change from BL at Day 2 | -2.1 (10.40) | -1.6 (8.82) | 2.8 (9.58)
  QTcF: Change from BL at Day 8 | -2.7 (9.54) | -1.0 (9.11) | 0.1 (8.51)

20. Secondary Outcome: Change From Baseline in Heart Rate Over Time, as Measured by Electrocardiogram
Description: A single 12-lead electrocardiogram (ECG) was obtained at the specified timepoints. To minimize variability in autonomic tone and heart rate, participants rested quietly and in a supine position for at least 5 minutes prior to recording the ECG. Blood draws, other procedures, activity, and environmental distractions (e.g., television, radio, conversation) were to be avoided during the pre-ECG resting period and between ECG recordings to minimize variability due to the effects of activity and stress on cardiac electrophysiology. Whenever possible, ECG tracings for each participant were to be obtained from the same type of machine throughout the study. The baseline value was defined as the last value recorded prior to the first dose in each treatment period. The normal reference range for heart rate was 50-100 beats per minute.
Time Frame: Baseline, and post-dose on Days 1, 2, and 8 of Periods 1-3 (up to 27 days)
Population: Safety Population: all participants who received at least one dose of study drug, grouped according to the treatment received.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C
Number analyzed (Participants) | 18 | 18 | 18
Beats per minute
  Baseline (BL) - Value at Visit | 62.3 (6.96) | 61.2 (6.71) | 62.4 (9.62)
  Change from BL at Day 1 | -2.9 (3.89) | -4.1 (6.53) | 0.5 (8.36)
  Change from BL at Day 2 | -1.0 (5.92) | -3.4 (6.03) | -4.6 (6.48)
  Change from BL at Day 8 | -0.2 (5.31) | 0.8 (4.71) | -0.9 (6.35)

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 14 days after the last dose of study drug (up to 41 days)
Arm/Group | GDC-9545 Tablet, Fasted: Treatment A | GDC-9545 Capsule, Fasted: Treatment B | GDC-9545 Capsule, Fed: Treatment C | Overall: Any GDC-9545 Treatment (A, B, or C)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 2/18 | 3/18 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GDC-9545 Tablet, Fasted: Treatment A (N=18) | GDC-9545 Capsule, Fasted: Treatment B (N=18) | GDC-9545 Capsule, Fed: Treatment C (N=18) | Overall: Any GDC-9545 Treatment (A, B, or C) (N=18)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Caution should be used when interpreting results from the statistical analyses conducted in this study because the sample size is not based on power calculations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the overall study. The Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT04274075/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-04): https://cdn.clinicaltrials.gov/large-docs/75/NCT04274075/SAP_001.pdf